CLINICAL TRIAL: NCT02423590
Title: A Phase II Randomised, Open-label Study of Gemcitabine/Carboplatin First-line Chemotherapy in Combination With or Without the Antisense Oligonucleotide Apatorsen (OGX-427) in Advanced Squamous Cell Lung Cancers
Brief Title: Study of Gemcitabine/Carboplatin First-line Chemotherapy +/- Apatorsen in Advanced Squamous Cell Lung Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009436QM
Record Dates: First submitted 2014-07-11; First posted 2015-04-22 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Squamous; Lung; Apatorsen
MeSH Terms: interventions — apatorsen; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine/Carboplatin (Active Comparator): Gemcitabine/carboplatin will be administered as standard 21-day treatment cycles according to normal clinical practice.
  * Gemcitabine will be given by 30 minute intravenous infusions on Day 1 and Day 8 of each 21-day Cycle.
  * On Day 1, carboplatin (AUC5) will be given by infusion over 30-60 minutes.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- Gemcitabine/carboplatin + Apatorsen (Experimental): * Apatorsen (OGX-427) will be administered as an intravenous infusion over 2 hours.
  * Apatorsen (OGX-427) treatment will begin with a loading dose period prior to the initiation of chemotherapy. Patients will receive three loading doses of 400 mg within a 9-day period with at least 48 hours between infusions and between the last loading dose infusion and Day 1 of initiating chemotherapy. Chemotherapy must be initiated within 7 calendar days once the last loading dose infusion has been completed.
  * Following the loading dose period, Apatorsen (OGX-427) will be given weekly at a dose of 400 mg by 2 hour intravenous infusions. On days when both chemotherapy and Apatorsen (OGX-427) are given, Apatorsen (OGX-427) should be given first followed by chemotherapy.
  Interventions: Drug: Apatorsen (OGX-427); Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Apatorsen (OGX-427) — Apatorsen (OGX-427) is a second generation antisense oligonucleotide designed to bind to Hsp27 mRNA
  Other Names: Apatorsen; OGX-427
  Arms: Gemcitabine/carboplatin + Apatorsen
Drug: Gemcitabine — Gemcitabine is an anti-cancer ("antineoplastic" or "cytotoxic") chemotherapy drug. Gemcitabine is classified as an antimetabolite
  Other Names: US Brand Name: Gemzar
Drug: Carboplatin — Carboplatin is an anticancer drug ("antineoplastic" or "cytotoxic") chemotherapy drug. Carboplatin is classified as an "alkylating agent."
  Other Names: Trade name: Paraplatin ®

SUMMARY:
This study is being carried out to see if a new drug called Apatorsen in combination with standard gemcitabine/carboplatin chemotherapy is effective in treating squamous cell lung cancer.

This study is part of a research project for collecting information about the effectiveness and safety of Apatorsen when used with gemcitabine/carboplatin chemotherapy. The main purpose of this study is to see if Apatorsen, when combined with gemcitabine/carboplatin, is an effective treatment for squamous cell lung cancer.

Recent research has found that a protein called Hsp27 can help cancer cells protect themselves against the effects of cancer treatments. Hsp27 is only found in some lung cancers but when it is present, cancer drugs might not work as well as they would without Hsp27 being present. Blocking the action of Hsp27 or removing Hsp27 from cancer cells with Apatorsen may slow down or stop the cancer growing. This study will therefore look at the relationship between the Hsp27 levels in tumour and blood and the effect of the treatment.

The development of Apatorsen is intended to provide a new treatment option for patients with cancer. Apatorsen may also make the cancer more sensitive to gemcitabine and carboplatin and so make this chemotherapy treatment more effective.

DETAILED DESCRIPTION:
This is an open-label, multicentre, 2-arm randomised phase II trial of gemcitabine/carboplatin + Apatorsen (OGX-427) versus gemcitabine/carboplatin alone in patients with previously untreated advanced squamous cell lung cancers. Patients will be randomised (1:1) to one of the two treatment arms:

* Gemcitabine/carboplatin
* Gemcitabine/carboplatin + Apatorsen (OGX-427)

Randomisation will be stratified by the following criteria:

* Stage (IIIB versus IV versus recurrent disease)
* Performance status (0 or 1 versus 2)

Gemcitabine/carboplatin chemotherapy will be continued for 4-6 cycles unless there is evidence of unacceptable toxicity, disease progression, or if the patient requests that study treatment be discontinued or to be withdrawn from the study. If chemotherapy is discontinued prior to disease progression, patients in the combination arm should be continued on Apatorsen (OGX-427) single agent therapy until disease progression unless there is evidence of unacceptable toxicity, patient withdrawal of consent or termination of the study, whichever occurs first. All patients will be followed for disease progression. Tumour evaluations will be performed before the initiation of treatment and every 6 weeks during and after completion of chemotherapy. Once disease progression is documented, patients will enter a Survival Follow-up Period during which data will be collected every two months regarding further cancer therapy, secondary malignancy and survival status. The study will also assess the relationship between the anticipated anti-tumour activity of the treatment regimen and biological characteristics of patients' tumours at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to admission to this study
2. Histological or cytological diagnosis of squamous non-small cell lung cancer. Patients with adenosquamous or mixed histology are not eligible for this study.
3. Stage IIIB disease that is unsuitable to radio-chemotherapy or Stage IV disease or recurrent NSCLC; recurrent disease must not be amenable to resection or radical radiotherapy with curative intent.
4. Patients must have:

   * at least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) OR
   * lytic or mixed (lytic + sclerotic) bone lesions in the absence of measurable disease as defined above
5. Willing to donate archival diagnostic tissue for translational research, if available.
6. Haematologic and biochemical indices within the ranges shown below. These measurements must be performed within one week prior to randomisation

   * ANC ≥1.5 x 109/L;, platelet count ≥100 x 109/L,
   * Serum creatinine < 1.5 times the upper limit of normal (ULN)
   * Bilirubin level < 1.5 X ULN
   * AST or ALT <3.0 X ULN or <5 X ULN in the presence of liver metastases
7. ECOG performance status 0-2
8. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant)
9. Male or Female aged ≥18 years

Exclusion Criteria:

1. Symptomatic CNS involvement or CNS involvement requiring steroid therapy; patients with treated brain metastases that are asymptomatic and have been clinically stable for 1 month will be eligible for protocol participation
2. Previous systemic treatment for lung cancer (exception for patients who have previously received immunotherapy without chemotherapy, and for patients with recurrent disease: adjuvant chemotherapy is allowed as long as this was finished at least 1 year prior to enrolment and did not contain gemcitabine)
3. Known tumour EGFR mutation, unless contraindication to EGFR-directed therapy
4. Known tumour ALK rearrangements, unless contraindication to Alk-directed therapy or Alk-directed therapy not available 1
5. Pre-existing sensory or motor polyneuropathy >Grade 2 according to NCI CTCAE
6. Significant cardiovascular disease, such as

   * History of myocardial infarction, acute coronary syndromes (including unstable angina), or history of coronary angioplasty/stenting/bypass grafting within past 6 months.
   * History of symptomatic congestive heart failure (CHF) New York Heart Association (NYHA) Classes III-IV.
   * Severe cardiac arrhythmia requiring medication or severe conduction abnormalities
   * Poorly controlled hypertension (resting diastolic blood pressure >115 mmHg)
   * Clinically significant valvular disease, cardiomegaly, ventricular hypertrophy, or cardiomyopathy
7. Active second malignancy (except non-melanomatous skin cancer): active secondary malignancy is defined as a current need for cancer therapy or a high possibility (>30%) of recurrence during the study.
8. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study entry.
9. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
10. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival as measured by investigator-assessed (using RECIST 1.1) progression-free survival | Date of patient randomisation to the date of first documented tumour progression (estimated 7.5 months) or death
  Progression-free survival, defined as the time from the date of randomisation to the date of first documented tumour progression based on investigator assessment (using RECIST 1.1) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Clinical Activity as measured by response rate (RECIST 1.1), change in tumour size, disease control rate, and duration of response of gemcitabine/carboplatin + Apatorsen relative to gemcitabine/carboplatin alone | At 12 weeks and 24 weeks post-randomisation until disease progression (estimated 7.5 months)
  Assess the clinical activity, as measured by response rate (RECIST 1.1), change in tumour size, disease control rate, and duration of response of gemcitabine/carboplatin + Apatorsen (OGX-427) relative to gemcitabine/carboplatin alone
Overall survival benefit of gemcitabine/carboplatin + Apatorsen relative to gemcitabine/carboplatin alone | Date of randomisation to date of death (expected average 12 months)
  Estimate the overall survival benefit of gemcitabine/carboplatin + Apatorsen (OGX-427) relative to gemcitabine/carboplatin alone
Clinical benefit as measured by investigator assessment using RECIST 1.1 | At 12 and 24 weeks post-randomisation
  Estimate the clinical benefit of gemcitabine/carboplatin + Apatorsen (OGX-427) relative to gemcitabine/carboplatin alone, as measured by investigator-assessed PFS rate at 12 and 24 weeks
Drug exposure measured as average dose per week | 4-6 cycles of treatment (12-18 weeks) and for apatorsen arm until disease progression (estimated 7.5 months)
  Evaluate drug exposure of gemcitabine/carboplatin + Apatorsen (OGX-427). Exposure is defined as average gemcitabine/carboplatin + Apatorsen (OGX-427) dose per week over whole treatment period.
  Gemcitabine/carboplatin chemotherapy will be continued for 6 cycles (each cycle is 21 days) unless there is evidence of unacceptable toxicity, disease progression, or if the patient requests that study treatment be discontinued or to be withdrawn from the study. If chemotherapy is discontinued prior to disease progression, patients in the combination arm should be continued on Apatorsen (OGX-427) single agent therapy until disease progression unless there is evidence of unacceptable toxicity, patient withdrawal of consent or termination of the study, whichever occurs first.
Compare the differences in health-related Quality of Life (HRQL) and symptoms for patients by treatment assignment as measured by the Functional Assessment of Cancer Therapy-Lung (FACT-L) scale, and the Euro-QOL 5D (EQ-5D) | Baseline, once every 3 weeks for 18 weeks and 4 weeks after last dose (estimated 8.8 months)
  Compare the differences in health-related quality of life (HRQL) and symptoms for patients by treatment assignment
Establish the safety and tolerability of gemcitabine/carboplatin + Apatorsen relative to gemcitabine/carboplatin alone | 3 weeks before treatment to 4 weeks after last dose (estimated 8.5 months)
  Establish the safety and tolerability of gemcitabine/carboplatin + apatorsen (OGX-427) relative to gemcitabine/carboplatin alone.
  This will include:
  * Incidence of serious adverse events
  * Incidence of grade 3 or higher adverse events (CTCAE, version 4.0)
  * Incidence of all adverse events of all grades
  * Incidence of infusion reactions and infusion-related adverse events
  * Adverse events leading to discontinuation of the study medication
  * Incidence of Grade 3 and 4 clinical laboratory results following study drug administration (CTCAE, version 4.0.3)

OTHER OUTCOMES:
Alterations in DNA and RNA | Baseline, day 1 of each cycle (each cycle is 21 days), every 3 weeks during maintenance and 4 weeks after last dose (estimated 8.5 months)
  Explore potential biomarkers that may help predict response to gemcitabine/carboplatin + Apatorsen (OGX-427) compared with gemcitabine/carboplatin alone.
Clinical Benefit, defined as number of patients with complete or partial response or stable disease maintained ≥24 weeks (as assessed by the site radiologist and/ or investigator, using RECIST 1.1) | 24 weeks until progression (estimated 7.5 months)
  Estimate the clinical benefit of chemotherapy + Apatorsen (OGX-427) relative to chemotherapy alone in patients with and without high Hsp27 expression in tumour tissue and by analysing the reduction of serum Hsp27 levels during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Prof., Study Chair — Queen Mary University London
Locations (20):
- United Kingdom (20):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Heart of England NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Velindre Cancer Centre, Cardiff
  - Colchester Hospital University NHs Foundation Trust, Colchester
  - Betsi Cadwaladr University Health Board, Denbighshire
  - NHS Tayside, Dundee
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - NHS Highland, Inverness
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Berkshire NHS Foundation Trust, Reading
  - Abertawe Bro Morgannwg University Health Board, Swansea
  - Weston Area Health NHS Trust, Weston-super-Mare
  - Yeovil District Hospital NHS Foundation Trust, Yeovil